CLINICAL TRIAL: NCT06836167
Title: + AGIL Barcelona: Integrated Care for Community-Dwelling Frail Older Adults
Brief Title: +AGIL Barcelona: Integrated Care for Community-Dwelling Frail Older Adults
Acronym: +AGIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc Sanitari Pere Virgili (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: +AGIL Barcelona; BDNS 604045 (Other Grant/Funding Number: trategic PPlan for Health Research and Innovation (PERIS))
Record Dates: First submitted 2025-01-13; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Older Adults; Healthy Aging
Keywords: frailty; older adults; Healthy Aging; integrated care; physical performance; intrinsic capacity
MeSH Terms: conditions — Frailty | interventions — Medication Review

STUDY DESIGN:
Intervention Model Description: Stepped-Wedge Cluster Randomized Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): During the adaptation phase of the program, all participating centers will begin by recruiting participants to the control group until they are transitioned to the recruitment of the intervention group. The control group will receive standard care plus educational materials focused on promoting a healthy lifestyle (videos or written materials, along with a weekly phone call to encourage viewing or address any questions). This is to avoid a bias related to the potential benefits of stricter follow-up in the intervention arm.
- Intervention (Experimental): The +AGIL program aligns with the World Health Organization's framework for Integrated Care for Older People (Ferrara MC et al., J Intern Med. 2023). It includes:
  1. Up to 10 weekly 1-hour group exercise sessions led by a physiotherapist, focusing on resistance, endurance, balance, and flexibility. Materials are adapted for low literacy or cognitive impairment, and Vivifrail® may be used to prevent frailty and falls.
  2. Non-pharmacological measures, such as guidance on the Mediterranean diet, screening for swallowing difficulties and cognitive decline, and advice on improving sleep.
  3. Support to reduce social isolation by connecting participants with community resources.
  4. A medication review to optimize treatments and deprescribe unnecessary drugs. The program has demonstrated significant improvements in physical performance and intrinsic capacity at three and six months, maintained through empowerment and ongoing connection to community resources.
  Interventions: Behavioral: exercise promotion; Drug: review medication; Behavioral: promoting healthy aging; Other: against social isolation

INTERVENTIONS:
Behavioral: exercise promotion — a) Up to 10 weekly 1-hour group sessions of multicomponent exercise guided by a physiotherapist, incorporating resistance, endurance, balance, and flexibility. Supported by materials adapted for low literacy or cognitive impairment, it empowers participants to maintain physical activity. Vivifrail may be used to prevent frailty and falls.
  Arms: Intervention
Drug: review medication — d) Comprehensive medication review for optimization and deprescribing. Results show significant improvements in physical performance and intrinsic capacity at three and six months, sustained through empowerment and community resource connections.
  Other Names: person centered review medication
  Arms: Intervention
Behavioral: promoting healthy aging — b) Non-pharmacological interventions, including nutritional guidance for a Mediterranean diet, dysphagia and cognitive impairment screening, and sleep hygiene counselling.
  Arms: Intervention
Other: against social isolation — Support against social isolation by activating community resources.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of the +AGIL Barcelona program in helping older adults improve their physical abilities and delay disability. It will also explore how to adapt and expand the program to different neighborhoods in Barcelona. The main questions it aims to answer are:

Does the +AGIL program improve physical abilities, as measured by a simple physical performance test (SPPB)? How well can the program be adapted and implemented in different community health centers? Researchers will conduct the study in three community health centers in Barcelona, following a stepped approach to gradually introduce the program at each site.

Participants will:

Participate in up to 10 weekly group exercise sessions led by a physiotherapist. Focus on strength, balance, flexibility, and endurance. Exercises will be tailored to individual needs and supported with easy-to-understand materials.

Receive advice on healthy habits like eating a Mediterranean diet, improving sleep, and managing swallowing or memory issues.

Get support to connect with local activities and resources to reduce loneliness and stay active, such as community centers or fitness programs.

Have their medications reviewed by healthcare professionals to ensure they are appropriate and safe.

The program will be personalized based on each participant's needs. This study will provide valuable information on implementing practical programs that help older adults stay healthy and independent.

DETAILED DESCRIPTION:
Population aging requires the implementation of sustained integrated strategies and programs to improve intrinsic capacity and delay disability in older adults. The +AGIL Barcelona program exemplifies a pragmatic, multicomponent intervention that effectively improves physical function by integrating health and community resources. This study aims to co-design, adapt, and scale up +AGIL to diverse socioeconomic areas in Barcelona, assessing its effectiveness and evaluating the process of progressive implementation.

Methods: Multicenter, pragmatic, Stepped-Wedge Cluster Randomized Trial, performed in three Primary Care Centers in Barcelona (PCCs), involving older adults screened as frail by the Gérontopôle Frailty Screening Tool (total sample size=396, 198 per arm). After a co-design phase to adapt the protocol to each local context, the intervention will be introduced sequentially at each site, according to a randomly determined schedule, until all PCCs are exposed. The intervention, previously piloted in a different PCC, is based on a Comprehensive Geriatric Assessment followed by a 10-week tailored boost multicomponent intervention aligned with the Integrated Care for Older People (ICOPE) framework of the World Health Organization - WHO - (physical exercise being the core element). After three months, continuity of activation is pursued through the integration of community resources (public or private gyms, civic centers etc). The primary outcome will be. The investigators designed a mixed-methods evaluation, measuring physical performance improvement using the Short Physical Performance Battery (SPPB) as the primary quantitative outcome, plus a qualitative assessment of participants' experience and program implementation.

Discussion: This study will provide relevant information on the implementation and impact of pragmatic, real-life interventions to improve intrinsic capacity and prevent disability in older adults.

ELIGIBILITY:
Inclusion Criteria:

* People aged 65 or older
* Presenting with suggestive signs of frailty according to the Gérontopôle Frailty Screening Test (GFST).
* Agree to participate and sign informed consent

Exclusion Criteria:

* Requirement for hospital admission or an estimated life expectancy of less than one year.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 396 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Physical performance | baseline, 3 months and 6 months
  measured using the Spanish-validated version of the Short Physical Performance Battery (SPPB). consistently with the previous demonstrator study, The SPPB includes sub-tests for balance, strength, and gait speed. Each sub-item is scored from 0 to 4 points, resulting in a maximum total score of 12, indicating optimal physical function. The SPPB is widely recognized as a predictor of disability in older adults. and serves as a primary indicator of frailty in this population. To assess the effectiveness of the +AGIL Barcelona program, we will use the total SPPB score and walking speed sub-item, which is also a strong predictor of adverse health outcomes in older populations.
  Scores range from 0 (worse) to 12 (maximum), values under 10 indicates frailty.

SECONDARY OUTCOMES:
Quality of life (QoL) | baseline, 3 months and 6 months
  will be measured using the EQ-5D-5L tool, which consists of two components:
  a) Health state description comprising 5 dimensions that assess mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on five levels: 1)No problems, 2) Slight problems, 3)Moderate problems, 4)Severe problems, and 5)Extreme problems
  The responses create a five-digit health profile (e.g., 11111 represents perfect health). These profiles can be converted into a single utility score using country-specific value sets.
  Maximum score (best health): 1.00 Minimum score (worst health): Typically less than 0 (values can go negative for states considered worse than death, depending on the value set used).
  B) a Visual Analog Scale for participants to provide an overall assessment of their health on a scale from 0 to 100.
  Maximun score 100: Best imaginable health, Minimum score 0: Worst imaginable health
Cognitive impairment | baseline, 3 months and 6 months
  will be screened using Mini-Cog®, a validated and quick tool that includes a 3-item recall test and a clock-drawing test. Scores range from 0 to 5 points, with a score below 3 indicating positive dementia screening.
Social engagement | baseline, 3 months and 6 months
  will be measured using the 6-item Lubben Social Network Scale (LSNS-6), with scores ranging from 0 to 30 (higher scores indicate greater social engagement).
Adherence to the Mediterranean diet | baseline, 3 months and 6 months
  will be assessed using the PREDIMED tool, whereas malnutrition risk will be measured using the MNA-Short Form (MNA-sf). An MNA-sf score of 12-14 points reflects normal nutritional status, 8-11 points suggests a risk of malnutrition, and 0-7 points suggest malnourishment.
Adverse events | baseline, 3 months and 6 months
  These include falls, fractures, cardiovascular events (such as angina, myocardial infarction, TIA, and stroke), hospital admissions, and mortality.
The total number of medications | baseline, 3 months and 6 months
  total number of medications, took from electronic health records and check it with participants and / or family

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Baro, MD, Principal Investigator — sbaro@perevirgili.cat
Locations (3):
- Spain (3):
  - Barceloneta - Primary Care Center, Barcelona
  - Larrad - Primary Care Center, Barcelona
  - Vila Olimpica - Primary Care Center, Barcelona

REFERENCES:
- [Background] Inzitari M, Perez LM, Enfedaque MB, Soto L, Diaz F, Gual N, Martin E, Orfila F, Mulero P, Ruiz R, Cesari M. Integrated primary and geriatric care for frail older adults in the community: Implementation of a complex intervention into real life. Eur J Intern Med. 2018 Oct;56:57-63. doi: 10.1016/j.ejim.2018.07.022. Epub 2018 Aug 23. PMID 30145055
- [Background] Perez LM, Enfedaque-Montes MB, Cesari M, Soto-Bagaria L, Gual N, Burbano MP, Tarazona-Santabalbina FJ, Casas RM, Diaz F, Martin E, Gomez A, Orfila F, Inzitari M. A Community Program of Integrated Care for Frail Older Adults: +AGIL Barcelona. J Nutr Health Aging. 2019;23(8):710-716. doi: 10.1007/s12603-019-1244-4. PMID 31560028
- [Background] Ferrara MC, Perez LM, Sole AR, Villa-Garcia L, Ars J, Soto-Bagaria L, Bellelli G, Cesari M, Enfedaque MB, Inzitari M. Sustained improvement of intrinsic capacity in community-dwelling older adults: The +AGIL Barcelona multidomain program. J Intern Med. 2023 Dec;294(6):730-742. doi: 10.1111/joim.13710. Epub 2023 Aug 21. PMID 37574781
- [Background] Canet-Velez O, Solis-Navarro L, Sitja-Rabert M, Perez LM, Roca J, Soto-Bagaria L, Torres-Castro R, Diaz-Gallego F, Vilaro J, Inzitari M. Experience, facilitators, and barriers to the implementation of a multicomponent programme in older people living in the community, +AGIL Barcelona: A qualitative study. Front Public Health. 2023 Mar 30;11:1161883. doi: 10.3389/fpubh.2023.1161883. eCollection 2023. PMID 37064681
- [Background] Arnal C, Perez LM, Soto L, Herrero AC, Ars J, Baro S, Diaz F, Abilla A, Enfedaque MB, Cesari M, Inzitari M. Impact on physical function of the +AGIL Barcelona program in community-dwelling older adults with cognitive impairment: an interventional cohort study. BMC Geriatr. 2023 Nov 13;23(1):736. doi: 10.1186/s12877-023-04292-4. PMID 37957601

DOCUMENTS (2):
  • Statistical Analysis Plan (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT06836167/SAP_000.pdf
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/67/NCT06836167/ICF_001.pdf